CLINICAL TRIAL: NCT06943248
Title: Effects of Image-Sand Play Therapy Versus Table Top Training Program With Weighted Cuffs on Visual Motor Integration in Children With Autism
Brief Title: Sand Play vs. Cuff Training: Visual-Motor Skills in Autism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/24/0750
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Sand play, Table-top training, Beery VMI
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A Randomized clinical trail performed, in which 30 children autism spectrum disorder with the age of 5-8 years will be taken after screening and meeting inclusion criteria. Children will be divided in two groups. Group A will perform Image-Sand Play Therapy Group had 12 week Image-Sand Play therapy, the one to one intervention provided once a week 30 min in each. Group B Table Top Training Program with Weighted Cuff Table Top training Program Duration: 12 week Patient perform each item 5 min with 1 min preparation between task . Pre values were taken at 1st week and then after 6th week mid values of interventions will be taken and post values of intervention will be taken after 12th week to measure the effect of both therapies .
Who Masked: Participant
Masking Description: Participants will be separate treatment protocol and possible efforts will be put to mask the both group about treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image-Sand Play Therapy (Experimental): Group A will perform Image-Sand Play Therapy Group had 12 week the one to one intervention provided once a week 30 min in each.
  Interventions: Other: Image-Sand Play Therapy
- Table Top Training Program with Weighted Cuff (Active Comparator): Table Top training Program Duration: 12 week Patient perform twice a week each item 5 min with 1 min preparation between task
  Interventions: Other: Table Top Training Program with Weighted Cuff

INTERVENTIONS:
Other: Image-Sand Play Therapy — Over the course of seven sessions, the child initially engaged in chaotic sandbox play, showing difficulty in altering or organizing his scenes. By the fourth session, he began experimenting with different symbols, including familiar TV characters. From the fifth session onward, his play gained structure, evolving into strategic battle scenarios involving animals, loggers, and castles. By the seventh session, hero figures emerged, and the therapist noted improved classroom behavior and cooperation, though social challenges with peers remained.
  Arms: Image-Sand Play Therapy
Other: Table Top Training Program with Weighted Cuff — Task include: Stacking cones Lift a cone with one hand and stack it on top of a fixed cone. (The difficulty level was controlled by using resistance bands of varying weights or instructing patients to sit or stand while performing the task.) Task Therapy Program Stacking 3 × 3 cm blocks Pick up blocks one at a time by using one hand and stack them. (The difficulty level was controlled by using resistance bands of varying weights.) Tailwind Use both hands to push the handles of an instrument up and down to the sounds of a metronome.
  (The difficulty level was controlled by varying the angle.) Pinch exerciser Take a pinch pin and put it on a rod. (The difficulty level was controlled by varying the resistance of the pinch pin (5 grades) and the diameter of the rod (3 grades).) O'Connor Tweezer Dexterity Test Pick up a pin (2.5 cm long) and put it in a 15 mm hole. (The difficulty level was controlled by using different tweezers.)
  Arms: Table Top Training Program with Weighted Cuff

SUMMARY:
This study compares Image-Sand Play Therapy and Tabletop Training with Weighted Cuffs for improving Visual-Motor Integration (VMI) in children with autism. A 12-week randomized controlled trial will be conducted at Tanzeem-ul-Nisan, Faisalabad. Beery VMI will assess outcomes. Data will be analyzed using SPSS-23. Non-probability conventional sampling will be used. Sessions occur twice weekly.

DETAILED DESCRIPTION:
This study compares the effectiveness of Image-Sand Play Therapy and Tabletop Training with Weighted Cuffs in improving Visual-Motor Integration (VMI) in children with autism.

Methods: A randomized controlled trial will be conducted with children diagnosed with autism from Tanzeem-ul-Nisan, Faisalabad. Participants will be randomly assigned to either intervention group. Both therapies will run for 12 weeks, with two sessions per week.

Image-Sand Play Therapy: Creative sand tray play guided by a therapist.

Tabletop Training: Structured tasks with weighted cuffs for proprioceptive input.

Assessment Tool: Beery VMI

Sampling: Non-probability conventional sampling

Data Analysis: SPSS version 23, using baseline, mid, and post-intervention scores to compare effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-8 yrs

  * A diagnosed by Autism
  * Guardian of child patients signed the informed consent
  * Both gender male and female

Exclusion Criteria:

* Complication of serious medical disease

  * Children and parents who cannot comply with the research
  * Surgical procedures performed in the year prior to the study
  * Poor medical conditions preventing participation

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Berry Visual Motor Integration | Baseline,4th week, 8th week and 12th week
  The Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI) is the gold standard for identifying difficulties in the coordination of visual and motor skills in adults and children. The Beery VMI based on the construction of test items, the Beery VMI has strong construct validity and strong predictive validity for academic outcomes. Visual motor Coordination takes around 10-15 min. The task is completed in three minutes. Excellent test-retest reliability (0.84-0.88)(16) Interrater reliability of (0.90 0.98). Internal consistency (0.81-0.82)
Nine Hole Peg Board | Baseline, 4th week ,8th week and 12th week
  The Nine Hole Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses(18, 19). Table (wooden or plastic): with 9 holes (diameter 10 mm, depth 15 mm) separated by 32 mm or 50 mm(20). Stick container: a square box (100 x 100 x 10 mm) separate from the boards or a shallow round container on top of the board. 9 pins (diameter 7 mm, length 32 mm)(21). Stopwatch Instruct the patient to remove the needles one by one from the container and insert them into the holes in the plate as quickly as possible, using only their hands. Ask the patient to remove the needles one by one from the holes and return them to the container. Excellent Test-retest reliability (ICC = 0.85). Excellent interrater reliability for the right hand (r = 0.984) and the left hand (r = 0.993) (22).

CONTACTS AND LOCATIONS:
Overall Officials: Hamna Faisal, MA-PPT, Principal Investigator — Rihah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patil O, Kaple M. Sensory Processing Differences in Individuals With Autism Spectrum Disorder: A Narrative Review of Underlying Mechanisms and Sensory-Based Interventions. Cureus. 2023 Oct 31;15(10):e48020. doi: 10.7759/cureus.48020. eCollection 2023 Oct. PMID 38034138